CLINICAL TRIAL: NCT01896687
Title: A Pilot Randomized Trial of Scrambler Therapy or Sham Treatment for Persistent Nonspecific Low Back Pain
Brief Title: Trial of Scrambler Therapy or Sham Treatment for Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM20002340; SCRA-LBP (Other: VCU)
Record Dates: First submitted 2013-05-13; First posted 2013-07-11 (Estimated); Results first posted 2014-09-15 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Low Back Pain
Keywords: nonspecific low back pain; chronic low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Scrambler therapy (Experimental): Scrambler therapy applied to region of low back pain for 30 minutes x 10 days
  Interventions: Device: Scrambler
- Sham Scrambler treatment (Sham Comparator): Sham treatment applied to region above low back pain at nontherapeutic dose for 30 minutes x 10 days
  Interventions: Device: Scrambler

INTERVENTIONS:
Device: Scrambler — Electrotherapy
  Other Names: Calmare

SUMMARY:
This pilot study will evaluate Scrambler therapy and Sham treatment on levels of low back pain, pain sensitivity and mRNA expression of pain sensitivity candidate genes.

DETAILED DESCRIPTION:
This pilot study will evaluate the feasibility of the experimental protocol and provide sufficient pilot data to estimate statistical power and sample size requirements. The study will include 30 individuals (15 per group) diagnosed with persistent low back pain who will receive a standard protocol of Scrambler therapy or sham treatment. Participant data will include subjective measures of low back pain, pain sensitivity using quantitative sensory testing, and mRNA expression levels of pain sensitivity candidate genes at baseline (prior to treatment) and 1 and 3 weeks post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* be 18-50 years of age
* diagnosed with persistent nonspecific LBP
* comprehend English

Exclusion Criteria:

* <18 or >50 years of age
* chronic pain at another site or associated with a painful condition
* pregnant or within 3 months post-partum
* implanted drug delivery system
* heart stents or metal implants such as pacemakers, automatic defibrillator, aneurysm clips, vena cave slips, or skull plates
* history of myocardial infarction or ischemic heart disease within the past six months
* history of epilepsy
* skin conditions such as open sores that would prevent proper application of electrodes

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Starkweather, PhD, ACNP-BC, Principal Investigator — Virginia Commonwealth University School of Nursing
Locations (1):
- Virginia Commonwealth University School of Nursing, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Starkweather AR, Coyne P, Lyon DE, Elswick RK Jr, An K, Sturgill J. Decreased low back pain intensity and differential gene expression following Calmare(R): results from a double-blinded randomized sham-controlled study. Res Nurs Health. 2015 Feb;38(1):29-38. doi: 10.1002/nur.21632. Epub 2015 Jan 8. PMID 25572279

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Scrambler Therapy | Sham Scrambler Treatment
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Scrambler Therapy | Sham Scrambler Treatment | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 7 | 4 | 11
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Worst Low Back Pain Score
Description: Low back pain will be measured by the Brief Pain Inventory (BPI). The BPI assesses the severity of pain, location of pain, pain medications, amount of pain relief in the past 24 hours and the past week, and the impact of pain on daily functions. For this study, the worst pain score will be used in the analysis. The worst pain score is rated from "0" meaning no pain to "10" meaning pain as bad as you can imagine.
Time Frame: baseline to 3 weeks post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scrambler Therapy | Sham Scrambler Treatment
Number analyzed (Participants) | 15 | 15
units on a scale
  Baseline Mean Worse Pain Score | 5.4 (2.1) | 4.9 (1.5)
  3-week post-treatment mean worst pain score | 3.2 (1.2) | 5.8 (1.7)
Statistical Analysis 1: Comparison: Scrambler Therapy vs Sham Scrambler Treatment; Test type: Superiority or Other; p < 0.001, ANOVA — The "worst" pain and interference scores as dependent variables, and time (baseline, 1-, and 3 week follow up visit), group (Calmare or Sham), and group by time interaction terms as the independent variable

ADVERSE EVENTS:
Time Frame: 1 month
Description: Information from standard questionnaires, investigator assessment, subjective measures of low back pain, and pain sensitivity levels using quantitative sensory testing will be documented at baseline (prior to treatment) and 1 and 3 weeks post-treatment. This information will be used as a means to assess for any serious or other adverse events.
Arm/Group | Scrambler Therapy | Sham Scrambler Treatment
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No